CLINICAL TRIAL: NCT05718102
Title: Pragmatic Trial to Enhance Quality Safety, and Patient Experience in COPD
Acronym: EQuiP COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PCORI-23668
Record Dates: First submitted 2023-01-25; First posted 2023-02-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Population Health Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist led (Active Comparator): Pharmacists will conduct population health management for patients with COPD
  Interventions: Other: Population-health management
- Pulmonologist led (Active Comparator): Pulmonologists will conduct population health management for patients with COPD
  Interventions: Other: Population-health management

INTERVENTIONS:
Other: Population-health management — Population-health management

SUMMARY:
Background: Over 26 million Americans have chronic obstructive pulmonary disease (COPD), which is the third leading cause of death in the United States. Unfortunately, few patients receive proven therapies and many receive therapies known to have safer alternatives. One major reason is the competing demands of primary care providers (PCPs) who manage 90% of patients with COPD. The research team has developed a population management approach where pulmonary specialists provide evidence-based recommendations as an E-consult with unsigned orders to PCPs. PCPs can then quickly review the E-consult and sign, modify, or discontinue these orders. The investigators found this intervention led to marked improvements in the quality-of-care delivered and patients' COPD-related quality-of-life. While promising, this approach is limited by a paucity of pulmonary providers nationwide. Clinical pharmacists are 20 times more prevalent as pulmonary specialists and some regions of VA (VISN 17, COPD Cares) have assigned clinical pharmacists a role in the management of patients with COPD. However, the relative effectiveness of pharmacist-led management is yet to be established.

Study Description: This study tests population management for COPD provided by pharmacists relative to pulmonary specialists. The investigators are conducting a cluster randomized clinical trial at five medical centers and their associated clinics within the Department of Veterans Affair. Study staff will randomize PCPs to population management conducted by either pulmonary specialists or pharmacists. Within PCPs' panels, study staff will use VA electronic health record to identify patients with evidence of COPD. Pulmonologists and pharmacists will review these patients and provide guideline-based recommendations to PCPs. Pulmonary specialists and pharmacists will then deliver evidence-based recommendations through E-consults coupled with unsigned orders for primary care providers to sign, modify or decline.

Outcomes: Investigators will assess if proactive, population management recommendations by clinical pharmacists and pulmonary specialists lead to non-inferior outcomes for patients with COPD. The primary outcome will be a composite endpoint of COPD exacerbation, pneumonia, hospitalization, or death six month after intervention. Secondary outcomes will include 1) the proportion of guideline recommended therapies received by patients, 2) COPD-related quality-of-life as measured by the Clinical COPD Questionnaire, and 3) PCP acceptance of recommendations, 4) each individual outcome within the primary composite endpoint above, and 5) patient- and caregiver-incurred costs.

ELIGIBILITY:
Inclusion Criteria:

* Participants may be PCP physicians and advance practice providers (APP) practicing at participating sites, and their patients who are diagnosed with or treated for COPD based on the following criteria:

  1. Recent discharge from hospital for COPD exacerbation
  2. Recent outpatient exacerbation (emergency room (ER), primary care)
  3. Received prescription for an inhaled corticosteroid (ICS) but does not meet criteria for ICS use
  4. Diagnosis of COPD and/or treatment and active smoker not receiving smoking cessation aide
  5. Treatment for COPD without evidence of spirometry within 10 years, or no airflow obstruction on existing spirometry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with COPD exacerbation, pneumonia, hospitalization, or Death (composite outcome) | 180 days after intervention

SECONDARY OUTCOMES:
COPD-related quality- of-life | 90 days after intervention
  Clinical COPD Questionnaire (CCQ). The CCQ includes 10 items encompassing three domains (symptoms, functional state, and mental state). Response options range from "never" to "almost all the time" and are scored from 0-to-6. The total score is calculated by the addition of each item divided by the total number of items, producing a range of scores between 0-6.
Proportion of patients with COPD exacerbation | 180 days after intervention
Proportion of patients with pneumonia | 180 days after intervention
Proportion of patients with hospitalization | 180 days after intervention
Proportion of patients with Death | 180 days after intervention
Quality of COPD care | 90 days after intervention
  Proportion of evidence-based practices received
Acceptance of Recommendations | 90 days after intervention
  Proportion of recommendations that are accepted by PCPs
Heterogeneity of treatment effect on primary and secondary outcomes by subgroup | 180 days after intervention
  Compare heterogeneity of treatment effect on primary and secondary outcomes by intervention priority/risk, age, race, sex, rurality, and multimorbidity.
Patient-incurred costs | 180 days after intervention
  Compare differences in incurred costs using electronic health record data and surveys to estimate costs for care related to COPD, pneumonia, and hospitalizations. These costs will include estimated costs for transportation, copays for visits and medications, and opportunity costs for time spent on care.
Caregiver-incurred costs | 180 days after intervention
  Compare differences in caregiver-incurred costs using electronic health record data and surveys to estimate costs incurred by caregivers for time spent accompanying patients to care related to COPD, pneumonia, and hospitalizations. These costs will include estimated costs for transportation and opportunity costs for time spent on care.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas M Donovan, MD, Principal Investigator — VA Puget Sound Health Care System; David H Au, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (5):
- United States (5):
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - Portland VA Medical Center, Portland, Oregon
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - VA Puget Sound Health Care System, Seattle, Washington
  - Mann-Grandstaff VA Medical Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will share a de-identified data set with the Patient-Centered Outcomes Research Institute-designated repository
Supporting Information: Study Protocol, SAP
Time Frame: 2028